CLINICAL TRIAL: NCT02982889
Title: A Phase 1 Randomized, Controlled, Double-Blind, Single Ascending Dose Safety and Pharmacokinetic/Pharmacodynamic Study in Healthy Adult Males After LIQ865 Injection
Brief Title: Single Ascending Dose Study of Two Liquidia Bupivacaine Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Liquidia Technologies, Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: LTI-111; 2016-002420-88 (EudraCT Number)
Record Dates: First submitted 2016-11-22; First posted 2016-12-06 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Acute Pain
Keywords: Analytical, Diagnostic,Therapeutic Technique and Equipment; Anesthesia and Analgesia
MeSH Terms: conditions — Acute Pain; Disease; Agnosia | interventions — Bupivacaine; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- LIQ865A bupivacaine formulation (Experimental): Liquidia's PRINT bupivacaine free base/PLGA (poly D,L-lactic-co-glycolic acid) suspension for subcutaneous injection at doses ranging from 150mg to 600mg
  Interventions: Drug: LIQ865A bupivacaine formulation; Drug: Diluent for LIQ865
- LIQ865B bupivacaine formulation (Experimental): Liquidia's PRINT bupivacaine free base suspension for subcutaneous injection at doses ranging from 150mg to 600mg
  Interventions: Drug: LIQ865B bupivacaine formulation; Drug: Diluent for LIQ865
- Diluent for LIQ865 (Placebo Comparator): Negative control for subcutaneous injection. Each subject will act as his own control, receiving a LIQ865 formulation subcutaneous injection in one calf, and a diluent subcutaneous injection in his other calf
  Interventions: Drug: LIQ865A bupivacaine formulation; Drug: LIQ865B bupivacaine formulation; Drug: Diluent for LIQ865
- 0.5% bupivacaine hydrochoride (Active Comparator): Positive control arm to be used with one of the LIQ865 cohorts, with each subject acting as his own positive control (i.e., one leg will receive subcutaneous injection of LIQ865A or LIQ865B, and the other leg will receive subcutaneous injection of 0.5% bupivacaine hydrochloride).
  Interventions: Drug: LIQ865A bupivacaine formulation; Drug: LIQ865B bupivacaine formulation; Drug: 0.5% bupivacaine hydrochoride

INTERVENTIONS:
Drug: LIQ865A bupivacaine formulation — single subcutaneous injection in medial calf
  Other Names: Marcaine; Marcaine Spinal; Sensorcaine; Sensorcaine-MPF; Sensorcaine-MPF Spinal; Marcaine HCl; Exparel
  Arms: 0.5% bupivacaine hydrochoride; Diluent for LIQ865; LIQ865A bupivacaine formulation
Drug: LIQ865B bupivacaine formulation — single subcutaneous injection in medial calf
  Other Names: Marcaine; Marcaine Spinal; Sensorcaine; Sensorcaine-MPF; Sensorcaine-MPF Spinal; Marcaine HCl; Exparel
  Arms: 0.5% bupivacaine hydrochoride; Diluent for LIQ865; LIQ865B bupivacaine formulation
Drug: Diluent for LIQ865 — Sterile diluent composed of 12.5mg/g sodium hyaluronate, 5.8mg/g sodium chloride, 1mg/g polysorbate 80, 6.1mg/g Tris base, in sterile water for injection - single subcutaneous injection
  Other Names: Hyaluronic Acid
  Arms: Diluent for LIQ865; LIQ865A bupivacaine formulation; LIQ865B bupivacaine formulation
Drug: 0.5% bupivacaine hydrochoride — single subcutaneous injection
  Other Names: Marcaine; Marcaine Spinal; Sensorcaine; Sensorcaine-MPF; Sensorcaine-MPF Spinal; Marcaine HCl; Exparel
  Arms: 0.5% bupivacaine hydrochoride

SUMMARY:
This study is designed to assess and characterize the safety and tolerability profile of LIQ865A and LIQ865B formulations compared to diluent or aqueous bupivacaine hydrochloride when infiltrated into a defined area of the medial calf, and to characterize bupivacaine plasma pharmacokinetic (PK) and pharmacodynamic (PD) profiles after a single dose of LIQ865A or LIQ865B, and to determine the individual plasma concentration/time curves and mean PK parameters of each product.

DETAILED DESCRIPTION:
Infiltration of an aqueous local anesthetic, for example, bupivacaine, into surgical sites at closure provides temporary analgesia, typically lasting up to 6 hours, and is one aspect of the multimodal approach to postsurgical analgesia or fast-track surgery. However, the limited duration of action of local anesthetics, even longer acting agents such as bupivacaine, result in patients who are likely to experience end of duration breakthrough pain before they are able to take or tolerate oral analgesics, thus necessitating the use of strong parenteral analgesics in the immediate postsurgical period. LIQ865A and LIQ865B are two distinct formulations of bupivacaine manufactured via Liquidia Technologies PRINT (Particle Replication In Non-wetting Templates), which Liquidia intends to pursue for product approval. Both formulations being tested have the potential for producing long-lasting control of post-surgical incisional pain.

ELIGIBILITY:
Inclusion Criteria:

* provide written informed consent prior to enrollment
* be a non-smoking male, American Society of Anesthesiologist (ASA) physical class 1 or 2
* have a BMI between 18.5 and 25 kg. inclusive, and a weight of at least 60 kg
* be willing and able to participate for the duration of the study
* be healthy on the basis of pre-study physical examination (PE), medical history review, vital signs, lab test results as specified in the protocol
* negative urine drug test results
* negative alcohol screening test
* negative antibody test results for hepatitis B, hepatitis C, and HIV

Exclusion Criteria:

* allergic to bupivacaine, or other amide local anesthetics, or the excipients in the LIQ865 formulations or the diluent
* has taken any concomitant medications or supplements for the 3 days prior to Day 0
* has been on blood thinner or medication affecting platelet formation for the 7 days prior to Day 0
* in the opinion of the investigator, is either a hyper or hypo-responder to screening sensitivity testing
* has a history of moderate or severe renal or hepatic impairment, moderate or severe active hepatic disease, or any other clinically significant medical condition that may preclude safe study participation
* has a clinically significant test result for any screening lab parameter
* has a history or ECG screening documentation of a clinically meaningful conduction abnormality
* has scarring, tattoos, infections, or other skin changes in the area of planned study medication injection
* has known neurological disease or dysfunction (central or peripheral) that may interfere with assessments
* is unable to adequately communicate with study staff, properly give informed consent, or otherwise comply with study procedures, particularly the ability to return for outpatient follow up visits
* has participated in another interventional clinical study (investigational or marketed product) within the 30 days prior to Day 0.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (AEs) | 30 days
  Safety assessments will include the incidence and severity of AEs during treatment and the follow-up period of the study

SECONDARY OUTCOMES:
Pharmacokinetic - Area under the plasma concentration curve from time zero to Day 5 | Timepoints (draws) at 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24 hours and 2, 3, 4, 5 days after treatment
Pharmacokinetic - Cmax (ng/mL) | Timepoints (draws) at 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24 hours and 2, 3, 4, 5 days after treatment
  Maximum plasma concentration over the entire sampling period, directly obtained from the experimental data of plasma concentration versus time curves, without interpolation.
Pharmacokinetic - Tmax (h) | Timepoints (draws) at 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24 hours and 2, 3, 4, 5 days after treatment
  Time to reach maximum plasma concentration
Pharmacokinetic - t1/2 (h) | Timepoints (draws) at 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24 hours and 2, 3, 4, 5 days after treatment
  Apparent terminal elimination half-life
Pharmacokinetic - CST1/2 (h) | Timepoints (draws) at 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24 hours and 2, 3, 4, 5 days after treatment
  Context-sensitive half-time measured from Tmax to time for plasma concentration to reach half of Cmax following study medication injection.
Pharmacodynamic Response - Pain intensity (Numeric Rating Scale) with Short Tonic Heat Stimulus (STHS) testing at various time points | 1, 2, 12, 24, 48, 72, 96, and 120 hours
  Testing done to calculate time-weighted Sum of Pain Intensity Differences (SPID) at the time points noted, compared to Baseline, and time specific SPID results
Pharmacodynamic Response - Change in Mechanical Pain Threshold (MPT) compared to Baseline using various time points | 12, 24, 48, 72, 96, and 120 hours
  Calculate the time-weighted sum of threshold differences (calculated as area-under-the-curve (AUC): AUC12, AUC24, AUC48, AUC72, AUC96, AUC120
Pharmacodynamic Response - Change in Heat Pain Threshold (HPT) compared to Baseline using various time points | 12, 24, 48, 72, 96, and 120 hours
  Calculate the time-weighted sum of threshold differences (calculated as area-under-the-curve (AUC): AUC12, AUC24, AUC48, AUC72, AUC96, AUC120
Pharmacodynamic Response - Change Mechanical Detection Threshold (MDT) compared to Baseline using various time points | 12, 24, 48, 72, 96, and 120 hours
  Calculate the time-weighted sum of threshold differences (calculated as area-under-the-curve (AUC): AUC12, AUC24, AUC48, AUC72, AUC96, AUC120
Pharmacodynamic Response - Change in Warmth Detection Threshold (WDT) compared to Baseline using various time points | 12, 24, 48, 72, 96, and 120 hours
  Calculate the time-weighted sum of threshold differences (calculated as area-under-the-curve (AUC): AUC12, AUC24, AUC48, AUC72, AUC96, AUC120
Pharmacodynamic Response - Change in Cold Detection Threshold (CDT) compared to Baseline using various time points | 12, 24, 48, 72, 96, and 120 hours
  Calculate the time-weighted sum of threshold differences (calculated as area-under-the-curve (AUC): AUC12, AUC24, AUC48, AUC72, AUC96, AUC120

CONTACTS AND LOCATIONS:
Overall Officials: Mads U Werner, MD, Principal Investigator — Multidisciplinary Pain Center, Rigshospitalet
Locations (1):
- DanTrial Aps, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No